CLINICAL TRIAL: NCT05363072
Title: Registry-based Non-interventional Analysis of Advanced/Metastatic Renal Carcinoma Treatment Patterns and Outcomes in the Hospital District of Southwest Finland.
Brief Title: A Study to Describe the Kidney Cancer Patient Population Treatment, and Results in the Hospital District of Southwest Finland.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061098; FIN-RCC-RWD (Other: Alias Study Number)
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-06

CONDITIONS: Renal Cell Cancer; Renal Cell Carcinoma; Cancer of Kidney; Cancer of the Kidney; Kidney Cancer; Kidney Neoplasms; Renal Cancer
Keywords: Advanced/ metastatic RCC (mRCC); Real World Evidence; Registry based study; Non-interventional study; Axitinib; Sunitinib; Pazopanib; Cabozantinib; Nivolumab; Sorafenib; Everolimus; Ipilimumab
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
The purpose of the study is to find out how patients with advanced kidney cancer have been treated in the hospital district of Southwest Finland over time.

ELIGIBILITY:
Inclusion Criteria:

For the characteristic group:

* Diagnosis of renal cell carcinoma (International Classification of Diseases 10th revision [ICD]-10:64) during 01 January 2010 and 31 December 2021

For the mRCC group:

* ICD-10 diagnosis code for metastasis (C77*-C79*), or
* American Joint Committee on Cancer (AJCC) stage 4, or AJCC stage data potentially not available for all patients
* Visit to oncologist (specialty code 65) with RCC as main diagnosis, or In Finland, the ICD-10 codes for metastatic disease are rarely used. In contrast, RCC patients visit oncologist, when and only when disease metastasises and therefore, the visit can be used as a proxy to a metastatic disease
* Initiation of treatment for mRCC

Exclusion Criteria:

For the characteristic group:

* Prevalent mRCC patients (i.e. diagnosis of metastatic RCC before 01 January 2010)
* Prevalent mRCC patients (i.e. diagnosis of RCC before 01 January 2010) if there is no records of metastatic disease during 2010-2021

For the mRCC group:

* Prevalent patients with mRCC (i.e. diagnosis of metastatic RCC before 01 January 2010)
* Patients without treatment for mRCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced/metastatic RCC and medical records available at the in the Hospital District of Southwest Finland (HDSF) HDSF registry
Sampling Method: Non-Probability Sample
Enrollment: 1112 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Finland, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Holsa O, Teittinen K, Anttalainen A, Ukkola-Vuoti L, Summanen M, Mattila KE. Observational study on the evolution of systemic treatments for advanced renal cell carcinoma in Southwest Finland between 2010 and 2021. Ther Adv Urol. 2023 Nov 5;15:17562872231206243. doi: 10.1177/17562872231206243. eCollection 2023 Jan-Dec. PMID 37941979
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4061098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included data from adult participants diagnosed with renal cell carcinoma (RCC) recorded in routine clinical practice and available in the medical records of the Hospital District of Southwest Finland (HDSF) data lake from January 2010 to December 2021.
Pre-assignment Details: A total of 1112 participants with incident RCC were included in the study. Data was evaluated over 1 month in this retrospective study.
Groups:
- All Participants With RCC: This study included participants diagnosed with RCC (local or metastatic) whose medical records were available at HDSF data lake irrespective of whether they received treatment. Participants were followed up from first record of RCC (index) until death, moved outside of HDSF or up to 31-Dec-2021.
Period: Overall Study
Arm/Group | All Participants With RCC
Started (All RCC participants) | 1112
Treated Metastatic RCC Participants (mRCC) | 191
Not Treated Metastatic RCC Participants | 145
Completed | 1112
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Arm/Group | All Participants With RCC
Number analyzed (Participants) | 1112
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Years
    All RCC participants | 69.3 (12.0)
    Treated mRCC participants: number analyzed (Participants) | 191
    Treated mRCC participants | 67.7 (8.5)
    Not-treated mRCC participants: number analyzed (Participants) | 145
    Not-treated mRCC participants | 74.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
  Participants
    All RCC participants: Female | 418
    All RCC participants: Male | 694
    Treated mRCC participants: number analyzed (Participants) | 191
    Treated mRCC participants: Female | 68
    Treated mRCC participants: Male | 123
    Not-treated mRCC participants: number analyzed (Participants) | 145
    Not-treated mRCC participants: Female | 57
    Not-treated mRCC participants: Male | 88
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Co-Diagnoses Before Index
Description: Number of participants according to co-diagnoses 3 years before participant's index were reported in this outcome measure. Index date was defined as the date of treatment initiation for mRCC. Co-diagnoses were based on International Classification of Diseases 10th revision (ICD-10) codes. One participant may have more than one co-diagnoses.
Time Frame: 3 years prior to index date
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included. This analysis was planned only in the treated mRCC participants.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With RCC
Number analyzed (Participants) | 191
Participants
  Infection | 139
  D41 Neoplasm of uncertain or unknown behavior of urinary organs | 45
  I10 Essential (primary) hypertension | 41
  R91 Abnormal findings on diagnostic imaging of lung | 26
  R31 Unspecified hematuria | 22
  E11 Non-insulin-dependent diabetes mellitus | 17
  E78 Disorders of lipoprotein metabolism and other lipidaemias | 16
  I48 Atrial fibrillation and flutter | 14
  G47 Sleep disorders | 13
  I26 Pulmonary embolism | 12
  H25 Senile cataract | 11
  J18 Pneumonia, organism unspecified | 11
  N40 Hyperplasia of prostate | 11
  R07 Pain in throat and chest | 11
  R10 Abdominal and pelvic pain | 11
  M17 Gonarthrosis [arthrosis of knee] | 10

2. Primary Outcome: Number of Participants According to Co-Diagnoses After Index
Description: Number of participants according to co-diagnoses up to 3 years after participant's index were reported in this outcome measure. Index date was defined as the date of treatment initiation for mRCC. Co-diagnoses were based on ICD-10 codes. One participant may have more than one co-diagnoses.
Time Frame: Up to 3 years after index date
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With RCC
Number analyzed (Participants) | 191
Participants
  Infection | 144
  I10 Essential (primary) hypertension | 32
  J18 Pneumonia, organism unspecified | 28
  R50 Fever of other and unknown origin | 28
  E11 Non-insulin-dependent diabetes mellitus | 15
  R10 Abdominal and pelvic pain | 15
  D41 Neoplasm of uncertain or unknown behavior of urinary organs | 14
  F43 Reaction to severe stress, and adjustment disorders | 14
  E87 Other disorders of fluid, electrolyte and acid-base balance | 13
  M54 Dorsalgia | 12
  R06 Abnormalities of breathing | 12
  R31 Unspecified hematuria | 12
  R53 Malaise and fatigue | 12
  G47 Sleep disorders | 11
  R91 Abnormal findings on diagnostic imaging of lung | 10

3. Primary Outcome: Body Mass Index (BMI)
Description: BMI of participants at index was reported in this outcome measure. Index date was defined as the date of treatment initiation for mRCC.
Time Frame: At index
Population: All eligible participants were included. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Kilogram per meter square
Arm/Group | All Participants With RCC
Number analyzed (Participants) | 1112
Kilogram per meter square
  All RCC participants | 27.3 (5.3)
  Treated mRCC participants: number analyzed (Participants) | 191
  Treated mRCC participants | 25.1 (4.3)
  Not-treated mRCC participants: number analyzed (Participants) | 145
  Not-treated mRCC participants | 26.5 (5.9)

4. Primary Outcome: Mean Outpatient Visits and Emergent Room Visits Per Patient Year
Description: The number of outpatient visits and emergency room (ER) visits per patient year for all contacts, disease-specific contacts and other contacts were reported in this outcome measure. All contacts included disease specific contacts and other contacts. Per patient year was defined as total sum of events divided by the total sum of follow-up length of the participants.
Time Frame: Up to maximum of 12 years (retrospective data collection of 1 month)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Mean (95% Confidence Interval); unit: Visits per patient year
Groups:
- Treated mRCC Participants: Participants with a diagnosis of advanced or metastatic RCC whose medical records were available at HDSF data lake and initiated treatment with sunitinib, pazopanib, cabozantinib, ipilimumab, nivolumab were included. Participants were followed up until death, moved outside of HDSF or end of study (31-Dec-2021).
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Visits per patient year
  Outpatient visits: All contacts | 29.37 [26.46 to 32.64]
  Outpatient visits: Disease-specific | 19.29 [17.36 to 21.52]
  Outpatient visits: Other contacts | 10.07 [8.13 to 12.3]
  ER visits: All contacts | 0.28 [0.19 to 0.38]
  ER visits: Disease-specific | 0.15 [0.09 to 0.21]
  ER visits: Other contacts | 0.14 [0.08 to 0.2]

5. Primary Outcome: Mean Number of Hospitalizations Per Patient Year
Description: The number of hospitalization visits per patient year for all contacts, disease-specific contacts and other contacts were reported in this outcome measure. All contacts included disease specific contacts and other contacts. Per patient year was defined as total sum of events divided by the total sum of follow-up length of the participants.
Time Frame: Up to maximum of 12 years (retrospective data collection of 1 month)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Mean (95% Confidence Interval); unit: Hospitalizations per patient year
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Hospitalizations per patient year
  All contacts | 1.25 [1.02 to 1.53]
  Disease-specific | 0.55 [0.43 to 0.7]
  Other contacts | 0.7 [0.56 to 0.87]

6. Primary Outcome: Mean Number of Procedures and Surgeries Per Patient Year
Description: Number of procedures and surgeries per patient year were reported in this outcome measure. Per patient year was defined as total sum of events divided by the total sum of follow-up length of the participants.
Time Frame: Up to maximum of 12 years (retrospective data collection of 1 month)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Mean (95% Confidence Interval); unit: Events per patient year
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Events per patient year
  Procedure: All contacts | 10.82 [9.5 to 12.42]
  Surgeries: All contacts | 0.77 [0.58 to 0.98]

7. Primary Outcome: Number of Participants According to Treatment
Description: Number of participants receiving each treatment per treatment line were reported in this outcome measure.
Time Frame: From initiation of treatment until death, moved outside of HDSF or end of study (maximum up to 12 years)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Participants
  1st line: Cabozantinib | 25
  1st line: Ipilimumab, Nivolumab | 8
  1st line: Other | 5
  1st line: Pazopanib | 24
  1st line: Sunitinib | 129
  2nd line: Axitinib | 21
  2nd line: Cabozantinib | 24
  2nd line: Everolimus | 15
  2nd line: Nivolumab | 12
  2nd line: Other | 0
  2nd line: Pazopanib | 22
  2nd line: Sorafenib | 9
  2nd line: Sunitinib | 6
  3rd line: Axitinib | 6
  3rd line: Cabozantinib | 8
  3rd line: Everolimus | 19
  3rd line: Nivolumab | 5
  3rd line: Pazopanib | 10
  3rd line: Sunitinib | 7

8. Primary Outcome: Number of Participants According to Treatment Per Treatment Line Between 2010 to 2017
Description: Number of participants according to treatment per treatment line between 2010 to 2017 were reported in this outcome measure.
Time Frame: Anytime between January 2010 to December 2017 (maximum up to 8 years)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Participants
  1st line: Other | 0
  1st line: Pazopanib | 19
  1st line: Sunitinib | 86
  2nd line: Axitinib | 18
  2nd line: Cabozantinib | 5
  2nd line: Everolimus | 12
  2nd line: Other | 0
  2nd line: Pazopanib | 18
  2nd line: Sorafenib | 9
  3rd line: Axitinib | 6
  3rd line: Everolimus | 12
  3rd line: Other | 5
  3rd line: Pazopanib | 9
  3rd line: Sunitinib | 5

9. Primary Outcome: Number of Participants According to Treatment Per Treatment Line Between 2018 to 2021
Description: Number of participants according to treatment per treatment line between 2018 to 2021 were reported in this outcome measure.
Time Frame: Anytime between January 2018 to December 2021 (maximum up to 4 years)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Participants
  1st line: Cabozantinib | 25
  1st line: Ipilimumab, Nivolumab | 8
  1st line: Other | 0
  1st line: Pazopanib | 5
  1st line: Sunitinib | 43
  2nd line: Cabozantinib | 19
  2nd line: Nivolumab | 10
  2nd line: Other | 16
  3rd line: Cabozantinib | 5
  3rd line: Everolimus | 7
  3rd line: Other | 6

10. Primary Outcome: Mean Number of Laboratory Days Per Patient Year
Description: Number of laboratory days per patient year were reported in this outcome measure. Per patient year was defined as total sum of events divided by the total sum of follow-up length of the participants.
Time Frame: Up to maximum of 12 years (retrospective data collection of 1 month)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Mean (95% Confidence Interval); unit: Days per patient year
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Days per patient year | 21.85 [19.95 to 24.04]

11. Primary Outcome: Mean Number of Laboratory Days Per Patient Year Stratified by International Metastatic Database Consortium (IMDC) Risk Category
Description: Number of laboratory days per patient year stratified by IMDC risk category were reported in this outcome measure. IMDC risk category included Score 0= favorable risk, no missing values allowed; Score 1-2= intermediate risk, total score=1: maximum 1 risk factor can have missing value, total score=2: no missing values allowed; Score 3-6= poor risk, maximum 3 risk factors allowed to have missing values; Unknown risk= when none of the above risk categories could be assigned. Per patient year was defined as total sum of events divided by the total sum of follow-up length of the participants.
Time Frame: Up to maximum of 12 years (retrospective data collection of 1 month)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Mean (95% Confidence Interval); unit: Days per patient year
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Days per patient year
  IMDC 0: number analyzed (Participants) | 15
  IMDC 0 | 21.46 [18.22 to 25.05]
  IMDC 1-2: number analyzed (Participants) | 81
  IMDC 1-2 | 20.26 [17.92 to 23.13]
  IMDC 3+: number analyzed (Participants) | 74
  IMDC 3+ | 28.26 [22.75 to 34.54]
  IMDC Unknown: number analyzed (Participants) | 21
  IMDC Unknown | 19.71 [16.22 to 26.77]

12. Primary Outcome: Number of Participants Classified According to Karnofsky Performance Status (KPS) Stratified by IMDC Risk Category
Description: KPS:used for rating activities of daily living on 11-step scale from 0-100,higher score=participant better able to carry daily activities.Score:100=normal no complaints;no disease evidence,90=able to carry normal activity;minor signs/symptoms of disease,80=normal activity with effort;some signs/symptoms, 70=cares for self;unable to carry normal activity,60=required occasional assistance,able to care for personal needs,50=required considerable assistance & frequent medical care,40=disabled;required special care/assistance,30=severely disabled;hospital admission indicated;20=very sick;hospital admission necessary,10=moribund & 0=dead.IMDC risk category:0=favorable risk,no missing values allowed;1-2=intermediate risk,total score=1:max 1 risk factor could have missing value,total score=2:no missing values allowed;3-6=poor risk,max 3 risk factors allowed to have missing values; Unknown=none of the above risk categories could be assigned.Index date=date of treatment initiation for mRCC.
Time Frame: At index
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With RCC
Number analyzed (Participants) | 191
Participants
  KPS: 10-40; IMDC 0 | 0
  KPS: 10-40; IMDC 1-2 | 0
  KPS: 10-40; IMDC 3+ | 8
  KPS: 10-40; IMDC unknown | 0
  KPS: 50-60; IMDC 0 | 0
  KPS: 50-60; IMDC 1-2 | 17
  KPS: 50-60; IMDC 3+ | 29
  KPS: 50-60; IMDC unknown | 5
  KPS: 70-80; IMDC 0 | 10
  KPS: 70-80; IMDC 1-2 | 48
  KPS: 70-80; IMDC 3+ | 34
  KPS: 70-80; IMDC unknown | 10
  KPS: 90-100; IMDC 0 | 0
  KPS: 90-100; IMDC 1-2 | 10
  KPS: 90-100; IMDC 3+ | 0
  KPS: 90-100; IMDC unknown | 0
  Missing; IMDC 0 | 0
  Missing; IMDC 1-2 | 0
  Missing; IMDC 3+ | 0
  Missing; IMDC unknown | 0

13. Primary Outcome: Number of Participants Classified According to Pathological Diagnosis (PAD) Histology
Description: Number of participants classified according to PAD were reported in this outcome measure. Histology included chromophobe renal cell carcinoma, clear cell renal cell carcinoma, oncocytoma renal cell carcinoma, papillary renal cell carcinoma, other (chromophobe, oncocytoma, and papillary renal cell carcinoma included if not reported separately) and missing. Index date was defined as the date of treatment initiation for mRCC.
Time Frame: At index
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants With RCC
Number analyzed (Participants) | 1112
Participants
  RCC participants: Chromophobe renal cell carcinoma | 41
  RCC participants: Clear cell renal cell carcinoma | 597
  RCC participants: Oncocytoma renal cell carcinoma | 27
  RCC participants: Papillary renal cell carcinoma | 105
  RCC participants: Other | 0
  RCC participants: Missing | 342
  Treated mRCC participants: Chromophobe renal cell carcinoma: number analyzed (Participants) | 191
  Treated mRCC participants: Chromophobe renal cell carcinoma | 0
  Treated mRCC participants: Clear cell renal cell carcinoma: number analyzed (Participants) | 191
  Treated mRCC participants: Clear cell renal cell carcinoma | 115
  Treated mRCC participants: Oncocytoma renal cell carcinoma: number analyzed (Participants) | 191
  Treated mRCC participants: Oncocytoma renal cell carcinoma | 0
  Treated mRCC participants: Papillary renal cell carcinoma: number analyzed (Participants) | 191
  Treated mRCC participants: Papillary renal cell carcinoma | 0
  Treated mRCC participants: Other: number analyzed (Participants) | 191
  Treated mRCC participants: Other | 11
  Treated mRCC participants: Missing: number analyzed (Participants) | 191
  Treated mRCC participants: Missing | 65
  Non-treated mRCC participants: Chromophobe renal cell carcinoma: number analyzed (Participants) | 145
  Non-treated mRCC participants: Chromophobe renal cell carcinoma | 0
  Non-treated mRCC participants: Clear cell renal cell carcinoma: number analyzed (Participants) | 145
  Non-treated mRCC participants: Clear cell renal cell carcinoma | 65
  Non-treated mRCC participants: Oncocytoma renal cell carcinoma: number analyzed (Participants) | 145
  Non-treated mRCC participants: Oncocytoma renal cell carcinoma | 0
  Non-treated mRCC participants: Papillary renal cell carcinoma: number analyzed (Participants) | 145
  Non-treated mRCC participants: Papillary renal cell carcinoma | 0
  Non-treated mRCC participants: Other: number analyzed (Participants) | 145
  Non-treated mRCC participants: Other | 8
  Non-treated mRCC participants: Missing: number analyzed (Participants) | 145
  Non-treated mRCC participants: Missing | 72

14. Other Pre Specified Outcome: Overall Survival
Description: Overall Survival was defined as the time from index (start of each treatment line) until death due to any cause or end of study. Overall survival according to treatment lines (1, 2 or 3) was presented in this outcome measure.
Time Frame: From index until death due to any cause or end of study (maximum up to 12 years)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Months
  Treatment line 1 | 21.4 [15.4 to 25.2]
  Treatment line 2: number analyzed (Participants) | 111
  Treatment line 2 | 14.9 [9.6 to 19.6]
  Treatment line 3: number analyzed (Participants) | 54
  Treatment line 3 | 13.8 [8.7 to 21.7]

15. Other Pre Specified Outcome: Time to Next Treatment (TTNT)
Description: Time to next treatment (TTNT) was defined as the interval between the start of current treatment and the start of the next-line treatment or death or end of study. Kaplan-Meier method was used for analysis. TTNT according to treatment lines were presented in this outcome measure.
Time Frame: From start of current treatment to date of next line treatment or death or end of study (maximum up to 12 years)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Months
  Treatment line 1 | 9.3 [7.5 to 11.1]
  Treatment line 2: number analyzed (Participants) | 111
  Treatment line 2 | 7.7 [3.9 to 12.3]
  Treatment line 3: number analyzed (Participants) | 54
  Treatment line 3 | 7.3 [5.1 to 8.6]

16. Other Pre Specified Outcome: Number of Participants Classified According to IMDC Risk Group Status at Initiation of Treatment
Description: Number of participants classified according to IMDC risk group status at initiation of treatment were reported in this outcome measure. IMDC risk category included score 0= favorable risk, no missing values allowed; score 1-2= Intermediate risk, total score=1: maximum 1 risk factor can have missing value, total score=2: no missing values allowed; Score 3-6= Poor risk, maximum 3 risk factors allowed to have missing values; Unknown risk= when none of the above risk categories could be assigned. Index date was defined as the date of treatment initiation for mRCC.
Time Frame: At index
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Participants
  IMDC 0 | 15
  IMDC 1-2 | 81
  IMDC 3+ | 74
  IMDC Unknown | 21

17. Other Pre Specified Outcome: Mean Absolute Costs Associated With Healthcare Resource Utilization
Description: Absolute costs associated with healthcare resource utilization for all contacts, disease-specific contacts and other contacts was reported in this outcome measure. All contacts included ER visits, hospitalizations, and outpatient contacts.
Time Frame: Up to maximum of 12 years (retrospective data collection of 1 month)
Population: All eligible advanced/metastatic RCC participants who initiated treatment for mRCC were included.
Measure: Mean (95% Confidence Interval); unit: Euros per patient year
Arm/Group | Treated mRCC Participants
Number analyzed (Participants) | 191
Euros per patient year
  All contacts | 15,473.75 [13,722.39 to 17,478.22]
  Disease-specific contacts | 9,114.95 [8,169.87 to 10,222.87]
  Other contacts | 6,358.79 [5,218.05 to 7,718.64]

ADVERSE EVENTS:
Time Frame: For all-cause mortality: From index until death due to any cause or end of study (maximum up to 12 years); For adverse events: not applicable as adverse events were not collected during the study.
Description: This observational retrospective study retrieved data from medical records and the data existed as unstructured data. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, minimum criteria for reporting an adverse event could not be met, hence adverse events were not collected and reported. All-cause mortality was only collected for treated mRCC participants.
Arm/Group | Treated mRCC Participants
All-Cause Mortality (participants affected / at risk) | 100/191
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT05363072/Prot_SAP_000.pdf